CLINICAL TRIAL: NCT05465044
Title: Incremental Hemodialysis for Veterans in the First Year of Dialysis (IncHVets): A Pragmatic, Multi-Center, Randomized Controlled Trial
Brief Title: Incremental Hemodialysis for Veterans in the First Year of Dialysis (IncHVets)
Acronym: INCHVETS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEPH-003-21F; CX002382 (Other: V A ORD CSRD); NEPH-003-21F (Other: VA ORD)
Record Dates: First submitted 2022-07-08; First posted 2022-07-19 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Chronic Kidney Disease (CKD) Stage 5; Kidney Dysfunction Requiring Dialysis (KDRD); Dialysis Dependency
Keywords: chronic kidney disease (CKD); Residual kidney function (RKF); Uremia; End-stage Renal Disease (ESRD); Hemodialysis; Dialysis adequacy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Uremia; Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized controlled trial (RCT)
Who Masked: Outcomes Assessor
Masking Description: Assessors blinded to the study intervention will interview patients using computer-adapted telephone interviewing for the main outcome measure (SF36 PCS)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Twice-Weekly Hemodialysis (Experimental): Twice-weekly hemodialysis with incremental crossover to thrice-weekly hemodialysis as indicated
  Interventions: Other: Twice-weekly hemodialysis with incremental crossover to thrice-weekly schedule
- Thrice-Weekly Hemodialysis (Placebo Comparator): Outright thrice-weekly hemodialysis without option to switch to less frequent dialysis schedule
  Interventions: Other: Thrice-Weekly Hemodialysis

INTERVENTIONS:
Other: Twice-weekly hemodialysis with incremental crossover to thrice-weekly schedule — 50% of the eligible participants will be assigned to twice-weekly hemodialysis for up to 12 months with incremental crossover to thrice-weekly hemodialysis as indicated.
  Arms: Twice-Weekly Hemodialysis
Other: Thrice-Weekly Hemodialysis — 50% of the eligible participants will be assigned to outright thrice-weekly hemodialysis, which will be continuation of the initial thrice-weekly schedule during the run-in period, without the option to switch to less frequent dialysis schedule representing the standard of care.
  Arms: Thrice-Weekly Hemodialysis

SUMMARY:
In this pragmatic clinical trial, which will dovetail with Veterans' routine outpatient dialysis clinic visits in six VA medical centers, the investigators will study 252 Veterans with kidney disease who need to start dialysis treatment. If a Veteran is eligible for the study by making enough residual urine, he/she will have a 50% chance to be offered the usual three-times-per-week dialysis vs. twice-per-week dialysis that is gradually increased to three-times per- week over one year. The investigators will compare health-related quality of life, how long residual kidney function lasts, and other measures including safety in these two groups. By conducting this study, the investigators hope to understand 1) whether starting dialysis with less frequency is safe, effective, and can help Veterans and their care-partners to better cope with dialysis, and 2) if incremental dialysis can result in major cost benefits to the VA health care system, thus allowing more patients to stay in VA dialysis clinics vs. being transferred to outside clinics.

DETAILED DESCRIPTION:
Each year approx. 12,000 Veterans with worsening kidney disease develop end-stage renal disease (ESRD) and initiate dialysis treatment. They comprise >10% of the US incident ESRD population. Dialysis is costly and associated with impaired health-related quality of life (HRQOL) and high mortality risk, especially in the first dialysis treatment year. Currently, starting treatment with outright full-dose thrice-weekly hemodialysis (HD) from the outset of therapy is the standard of care regardless of patients' residual kidney function (RKF) and regardless of patients' and care-partners' suffering and preferences. Although not currently the standard of care, evidence suggests that gradual or incremental dialysis transition using an initial twice-weekly HD may confer substantial benefits including more dialysis-free time, longer RKF preservation, less trauma to patients' organs including their dialysis vascular access, lower frequency of intradialytic hypotensive events, less post-dialysis fatigue, and reduced patient suffering. Hence, incremental dialysis transition may result in improved HRQOL through better physical function, less fatigue, more energy, and better patient satisfaction and life participation by mitigating the burden of excessive dialysis in day-to-day life and on employment. Pragmatic studies with immediate impact are needed to shift the focus of dialysis from abrupt thrice-weekly HD start to a safe and effective personalized dialysis regimen.

In this multi-site, pragmatic, 1:1 randomized controlled trial (RCT), parallel with Veterans' routine dialysis therapy, the investigators will test the safety and efficacy of an incremental HD protocol, compared to standard-of-care thrice-weekly HD, in Veterans who meet the eligibility criteria. The investigators plan to compare twice-weekly (incremental) with thrice-weekly (conventional) HD initiation in 252 Veterans, who will transition to maintenance HD therapy in six VA centers. Assessing quarterly for up to 12 months, the investigators will study HRQOL physical health score as the primary endpoint, as well as dialysis symptom index and energy/fatigue score as secondary endpoints. Additional secondary outcome measures to collect and examine quarterly include preservation of the RKF, dialysis adequacy, nutritional status, and serum level of Growth Differentiation Factor 15. Safety assessments will include mortality, dialysis withdrawals, ER visits, hospitalizations, hyperkalemia, and major adverse cardiovascular events. In a substudy of 112 participating Veterans in three VA centers, the investigators will additionally examine cardiac measures including left ventricular mass, as well as mid-arm muscle circumference and physical performance.

This pragmatic RCT addresses a major unmet need in those Veterans who initiate dialysis by focusing on improving HRQOL and preserving RKF, the two strongest predictors of survival and patients' satisfaction. The results of the study may enable more Veterans to receive therapy in a VA based dialysis center. The study could lead to a paradigm shift with immediate impact on kidney care in Veterans and in the broader population with ESRD. The study challenges the current standard of care of outright thrice weekly HD in the first year of dialysis therapy, during which patients suffering and mortality are the highest, and is less likely to be supported by for-profit dialysis providers given the perceived reduction in revenue if twice-weekly HD is to be implemented broadly.

ELIGIBILITY:
Inclusion Criteria:

* Adult Veterans diagnosed with ESRD and who will soon need chronic dialysis initiation or have initiated hemodialysis (HD) not longer than 8 weeks of the target randomization day in one of the six VA centers.
* Meeting the incremental dialysis eligibility criteria in Table 4* under the IncHVets Study Protocol.
* Willingness to undergo the randomly assigned modality of 2x/wk vs 3x/wk HD.
* Willingness to attend the baseline and quarterly study tests in the dialysis unit or via telehealth as determined by study staff, which will mostly be parallel to the routine dialysis clinic visits.
* Agreeable to receive monthly or more frequent reviews for and interviews, regardless of being assigned to the incremental or conventional dialysis group.
* As shown in Table 4 of the INCHVETS Study protocol under incremental dialysis criteria, eligible subjects must have a urine output >0.5 L/day and urea clearance (KRU) >3 ml/min and meet 5 or more of the 9 other incremental dialysis criteria , which are derived from the 2014 Incremental Dialysis Consensus paper (Kalantar-Zadeh et al. Twice-weekly and incremental hemodialysis treatment for initiation of kidney replacement therapy. Am J Kidney Dis. 2014 Aug;64(2):181-6. doi: 10.1053/j.ajkd.2014.04.019. PMID: 24840669 PMCID: PMC4111970)

Exclusion Criteria:

* Having a terminal illness with a life expectancy less than 6 months such as stage 4 metastatic cancer or having signed for hospice with life expectancy less than 6 months.
* A serum potassium level >6.0 mEq/L during the 4 weeks prior to the study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change over time in numeric scale of Health-Related Quality of Life (HRQOL) Physical Component Score (PCS) of SF36 questionnaire. | Change over 12 months based on measuring at baseline and at Month 3, 6, 9 and 12
  The primary endpoint under Aim 1 will be HRQOL Physical Component Score (PCS) measured by the SF36, assessed at baseline and Month 3, 6, 9 and 12. SF36 questionnaires will be administered by trained assessors blinded to the intervention assignment using computer adapted telephone interviewing for SF36. It is a numeric value from 0 (worse) to 100 (best HRQOL physical score).

SECONDARY OUTCOMES:
Change over time in numeric scale of SF36 Energy/Fatigue Subscale off SF36 HRQOL | Change over 12 months based on measuring at baseline and at Month 3, 6, 9 and 12
  This subscale of SF36 under Vitality domain captures patients' reported state of feeling fatigued vs. having energy under Aim 1 as secondary endpoint. It is a numeric value from 0 (worse) to 100 (best vitality).
Change over time in in numeric score of Dialysis Symptom Index (DSI) | Change over 12 months based on measuring at baseline and at Month 3, 6, 9 and 12
  The Dialysis Symptom Index (DSI) includes 30 items related to physical and emotional symptoms. The tool was developed for HD patients, has excellent internal consistency, test-retest reliability, group differences validity, which will be under Aim 1 as a secondary endpoint. It is a numeric value from 0 (least bothering symptoms) to 120 (worse bothering symptoms).
Change over time in residual urine output (UOP) in ml/day | Change over 12 months based on measuring at baseline and at Month 3, 6, 9 and 12
  Baseline and quarterly residual kidney function (RKF) data will be collected, and 24-hr urine volume and endogenous urea clearance (Kru) will be calculated under Aim 2. It is a numeric value in ml per day from none (no urine output) to 3,000 cc/day or higher urine output.
Change over time in numeric value of Total Dialysis Adequacy (KT/V, sum of dialysis and residual kidney urea clearance) | Change over 12 months based on measuring at baseline and at Month 3, 6, 9 and 12
  Baseline and quarterly residual kidney function (RKF) data will be collected, and 24-hr urine volume and endogenous urea clearance (Kru) will be calculated under Aim 2. Total Dialysis Adequacy, known as KT/V, is the sum of dialysis machine generated adequacy (kt/v) and residual kidney urea clearance in commensurate units to be able to add up, resulting in a numeric value that usually ranges from 0.5 (low adequacy) to 2.5 (high adequacy) but even lower and higher values can rarely be observed.
Change over time in numeric scale of Malnutrition-Inflammation Score (MIS) | Change over 12 months based on measuring at baseline and at Month 3, 6, 9 and 12
  The Malnutrition-Inflammation Score (MIS) is a validated tool for longitudinal nutritional assessment of patients with CKD to detect Protein-Energy Wasting (PEW). MIS is a user-friendly tool requiring several minutes to assess nutritional status based on 10 criteria including 7 components of the Subjective Global Assessment (SGA) as well as commensurate ranked values that are generated to represent predefined increments of body mass index and serum albumin and transferrin levels, with a uniform 4-point Likert scale ranging from 0 to 3 (least to most severe malnutrition) across all 10 components and an overall nutritional severity score between 0 (best nutritional status with no malnutrition) and 30 (worse nutritional status).
Change over time in Serum level of Growth Differentiation Factor 15 (GDF15) | Change over 12 months based on measuring at baseline and at Month 3, 6, 9 and 12
  Growth Differentiation Factor 15 (GDF15) (measured via ELISA, R&D systems Inc., Minneapolis, MN) is a TGF- superfamily protein that that acts upon the hypothalamus to reduce food intake and energy expenditure, and it is associated with anorexia, weight loss, lower lean body and fat mass, and decreased survival. In clinical studies of dialysis-associated PEW, higher GDF15 levels have been associated with worse body composition (i.e., lower levels of skeletal muscle and fat), poorer nutritional status, weight loss, and death. In the INCHVETS trial, GDF15 levels will be measured as a marker of PEW and nutritional status in the main study at baseline and quarterly as the only non routine laboratory test. In our dialysis patient studies, GDF15 levels has a mean 5.94 and SD of ±3.90 ng/mL, ranging from 1.58 to 39.8 ng/mL (You et al Cardiorenal Med. 2017; 7(2): 158-168. doi: 10.1159/000455907).

OTHER OUTCOMES:
Change over time in numeric scale of Short Physical Performance Battery (SPPB) | Change over 12 months based on measuring at baseline and at Month 6, and 12 in the sub-study of 112 participants
  In order to measure physical performance, coordinators will conduct the SPPB on HD days within minutes before HD commences at baseline and at Months 6 and 12. The SPPB tests 1) gait speed (faster of two timed, usual pace 15-foot walks), 2) balance (balance test measuring ability to stand with feet in side-by-side, semi-tandem, and tandem positions for 10 seconds), and 3) chair raises (timed series of five attempts to arise from a chair unassisted without use of arms), with each component ranging from 0 to 4, i.e., score 0-12; higher score indicates better functional performance.
Change over time in mid-arm muscle circumference (MAMC) in cm | Change over 12 months based on measuring at baseline and at Month 6, and 12 in the sub-study of 112 participants
  In the sub-study, this conveniently measured and calculated value will be assessed as an exploratory outcome derived from triceps skinfold and mid-arm circumference measurements under Aim 3. The MAMC ranges usually from 20 to 40 cm (highest representing more muscle mass).
Change over time in Left Ventricular (LV) mass | Over 12 months (from baseline and at Month 12) in the sub-study of 112 participants
  The left ventricular (LV) mass will be measured via post-HD 2D-echo as the Cardiovascular domain under Aim 4. This metric is assessed via echocardiogram, and larger LV mass and increase in value over time is associated with unfavorable status and clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Kamyar Kalantar-Zadeh, MD PhD, Principal Investigator — VA Long Beach Healthcare System, Long Beach, CA
Locations (6):
- United States (6):
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York
  - Memphis VA Medical Center, Memphis, TN, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: INCHVETS study updates and announcements will be posted here — http://www.INCHVETS.com